CLINICAL TRIAL: NCT01948271
Title: An Open-label Pilot Study to Assess the Safety and Efficacy of Trichuris Suis Ova for the Treatment of Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Efficacy Study of Trichuris Suis Ova to Treat Chronic Plaque Psoriasis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSOPSO13
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Psoriasis
Keywords: Psoriasis; Trichuris suis ova; T-lymphocytes
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TSO 7500 (Experimental): Subjects in this arm will receive doses of 7500 trichuris suis ova every two weeks, starting at the baseline visit, for a total of 8 doses.
  Interventions: Drug: Trichuris Suis Ova

INTERVENTIONS:
Drug: Trichuris Suis Ova — During the treatment phase, study drug will be provided in a liquid form and will be administered every 2 weeks, starting with the Baseline visit, through Week 14.
  Other Names: TSO 7500

SUMMARY:
The purpose of this research study is to better understand whether trichuris suis ova (TSO) ingested orally may be safe and effective in the treatment of psoriasis.

DETAILED DESCRIPTION:
This is an open-label study to assess the safety and efficacy of 16 weeks of treatment with 7500 trichuris suis ova (TSO 7500) given every 2 weeks (a total of 8 doses) for the treatment of moderate-to-severe, chronic, plaque-type psoriasis.

ELIGIBILITY:
Inclusion criteria:

1. Males or females, 18-75 years old
2. Diagnosis of stable plaque type psoriasis for at least 6 months prior to baseline
3. Baseline moderate to severe psoriasis, defined as:

   1. Psoriasis covering a body surface area (BSA) ≥10%;
   2. Physician's global assessment (PGA) ≥3, and;
   3. PASI ≥12
4. Must be in good health as judged by the PI, based on medical history, physical examination, and clinical laboratories
5. In the opinion of the PI, must be a candidate for systemic therapy or phototherapy of psoriasis
6. If a woman, before entry she must be one of the following:

   1. Postmenopausal, defined as 45 years of age with amenorrhea for at least 18 months, or >45 years of age with amenorrhea for >6 months and a serum follicle stimulating hormone (FSH) level >40 IU/mL, or surgically postmenopausal (bilateral oophorectomy)
   2. surgically sterile (have had a hysterectomy or tubal ligation or otherwise be incapable of pregnancy)
   3. If heterosexually active, practicing a highly effective method of birth control, including hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method (eg, condoms, diaphragm, or cervical cap, with spermicidal foam, cream, or gel), or male partner sterilization for the duration of their participation in the study and for 2 months after receiving the last administration of any study agent; or
   4. Not heterosexually active
7. Women of childbearing potential must have a negative pregnancy test (urine and serum) prior to randomization
8. Agree to avoid prolonged exposure to natural sunlight or tanning beds or phototherapy devices for the duration of the study
9. Agree to avoid any prohibited concomitant medications as detailed below for the duration of the study and for 4 weeks prior to baseline
10. Negative stool culture
11. Subject has the ability to provide informed consent
12. Subjects who are on inhaled or ophthalmic steroids are allowed

Exclusion Criteria:

1. Subjects with known history of intestinal parasitic infection, even if adequately treated, in the past 5 years
2. Subject received antibiotic, antifungal or antiparasitic medication in the last 2 weeks prior to Screening and/or would potentially require this during the study treatment period
3. Subject with history of drug or alcohol abuse within 6 months prior to screening
4. Subject with evidence of poor compliance with medical advice and instruction including diet or medication
5. Subject is unable or unwilling to swallow study medication suspension
6. Subject with a significant medical condition which puts the subject at risk for study participation and/or for any reason is considered by the Investigator to be an unsuitable candidate to receive TSO or is potentially put at risk by study procedures
7. Subjects who has participated in another clinical trial within 30 days of screening for this trial and/or any experimental treatment for this population
8. White blood cell count ≤3,000/mm3 (≤3.0 x 109/L) or ≥14,000/mm3 (≥14 x 109/L)
9. Platelet count ≤ 100,000/μL (≤100 x 109/L)
10. Serum creatinine >2 x upper limit of normal (ULN)
11. Aspartate or alanine aminotransferase >2 x ULN
12. Total bilirubin >2 mg/dL (34 μmol/L)
13. Hemoglobin < 9 g/dL
14. Subjects who are currently taking or have taken in the past 30 days, for any reason, any medication that, in the opinion of the investigator, suppressed the immune response. This may include but is not limited to systemic steroids, azathioprine, cyclosporine, tacrolimus, mycophenolate mofetil, mycophenolic acid, etanercept, adalimumab, infliximab, ustekinumab, cimzia, or any other biologic agent targeted to any cell or cytokine in the immune system.
15. Subjects who are refractory to 2 or more biological agent plaque psoriasis therapies due to lack of efficacy
16. Subjects currently taking or who have taken in the past 2 weeks, topical steroids
17. Subjects on a non-stable dose of vitamin D analog in the past 30 days
18. Subjects currently taking or who have taken in the past 30 days any medications likely to improve psoriasis and thus interfere with evaluation. This may include, in addition to the medications listed above, phototherapy, methotrexate, hydroxyurea, or acitretin
19. Subjects with a diagnosis of inflammatory bowel disease (ulcerative colitis or Crohn's disease) or of irritable bowel syndrome
20. Subjects with HIV-1/HIV-2 antibody, hepatitis B surface antigen, hepatitis C antibody
21. Subject received non-steroidal anti-inflammatory drugs within 2 weeks before Baseline visit for more than 3 consecutive days, except acetylsalicylic acid ≤350 mg/d which is allowed
22. Women who are intending to become pregnant or who are breastfeeding or planning to breastfeed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Physician's area and severity index (PASI) | Screening, baseline, weeks 2, 4, 6, 8, 10, 12, 14, and 16
  The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. PASI produces a numeric score that can range from 0 to 72 based on the body surface area of involvement and the severity of disease (induration, erythema and scale). A PASI-50 response is defined as ≥50% improvement in PASI score from baseline; PASI-75 and PASI-90 are similarly defined.

SECONDARY OUTCOMES:
Safety and tolerability | Screening, baseline, weeks 2, 4, 6, 8, 10, 12, 14, 16, 20, and 38
  Evaluated via the frequency and severity of adverse events, changes in physical examinations, stool studies (ova and parasites, culture, clostridium difficile toxin, and blood), clinical laboratories (liver function tests, creatine phosphokinase, complete metabolic profile, complete blood count), and vital signs (blood pressure, pulse and temperature).

CONTACTS AND LOCATIONS:
Overall Officials: Alice B Gottlieb, MD, PhD, Principal Investigator — Tufts Medical Center, Department of Dermatology
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrett JC, Hansoul S, Nicolae DL, Cho JH, Duerr RH, Rioux JD, Brant SR, Silverberg MS, Taylor KD, Barmada MM, Bitton A, Dassopoulos T, Datta LW, Green T, Griffiths AM, Kistner EO, Murtha MT, Regueiro MD, Rotter JI, Schumm LP, Steinhart AH, Targan SR, Xavier RJ; NIDDK IBD Genetics Consortium; Libioulle C, Sandor C, Lathrop M, Belaiche J, Dewit O, Gut I, Heath S, Laukens D, Mni M, Rutgeerts P, Van Gossum A, Zelenika D, Franchimont D, Hugot JP, de Vos M, Vermeire S, Louis E; Belgian-French IBD Consortium; Wellcome Trust Case Control Consortium; Cardon LR, Anderson CA, Drummond H, Nimmo E, Ahmad T, Prescott NJ, Onnie CM, Fisher SA, Marchini J, Ghori J, Bumpstead S, Gwilliam R, Tremelling M, Deloukas P, Mansfield J, Jewell D, Satsangi J, Mathew CG, Parkes M, Georges M, Daly MJ. Genome-wide association defines more than 30 distinct susceptibility loci for Crohn's disease. Nat Genet. 2008 Aug;40(8):955-62. doi: 10.1038/ng.175. Epub 2008 Jun 29. PMID 18587394
- [Background] Baumgart DC, Sandborn WJ. Inflammatory bowel disease: clinical aspects and established and evolving therapies. Lancet. 2007 May 12;369(9573):1641-57. doi: 10.1016/S0140-6736(07)60751-X. PMID 17499606
- [Background] Crohn BB, Ginzburg L, Oppenheimer GD. Regional ileitis: a pathologic and clinical entity. 1932. Mt Sinai J Med. 2000 May;67(3):263-8. No abstract available. PMID 10828911
- [Background] Loftus EV Jr, Schoenfeld P, Sandborn WJ. The epidemiology and natural history of Crohn's disease in population-based patient cohorts from North America: a systematic review. Aliment Pharmacol Ther. 2002 Jan;16(1):51-60. doi: 10.1046/j.1365-2036.2002.01140.x. PMID 11856078